CLINICAL TRIAL: NCT02932787
Title: Effects of Installing Height-adjustable Workstations on Occupational Sitting Time and Workplace Productivity in Desk-based Workers
Brief Title: Effects of Installing Height-adjustable Workstations on Office Workers Workplace Sitting Time and Productivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Hallam University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SHU-AWS-RCT
Record Dates: First submitted 2016-09-23; First posted 2016-10-13 (Estimated); Results first posted 2020-04-28 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Workplace Inactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Height-adjustable workstation (Experimental): Participants received a height-adjustable workstation for four weeks
  Interventions: Device: Height-adjustable workstation
- Control (No Intervention)

INTERVENTIONS:
Device: Height-adjustable workstation
  Arms: Height-adjustable workstation

SUMMARY:
The purpose of this study was to look at the effects that height-adjustable workstations on occupational sitting time and workplace productivity in office workers. Participants workplace activity (sitting, standing and walking) and productivity was measured before the installation of the height-adjustable workstations. Workplace activity and productivity were then measured four weeks after the installation of height-adjustable workstations. The results were compared to a control group who received no intervention whilst the intervention had the height-adjustable workstations.

DETAILED DESCRIPTION:
Sedentary behaviour has been found to be ubiquitous within the workplace and due to the negative consequences of sedentary behaviour upon health, research has began to look at ways to reduce and interrupt sedentary behaviour.

Interventions that have introduced height-adjustable workstations into the workplace have been found to reduce sedentary behaviour. Some employees and employers are concerned that using height-adjustable workstations and trying to reduce workplace sedentary behaviour can lead to a loss of workplace productivity.

The present study looked at the effects of installing height-adjustable workstations on occupational sitting time and workplace productivity in desk-based workers. Workplace activity was measured objectively using ActivPal accelerometers and productivity was measured via self-report measures. Measurements took place at baseline and four weeks after receiving the height-adjustable workstation.

ELIGIBILITY:
Inclusion Criteria:

1. age 18 to 65 years,
2. working ≥0.6 full time equivalents,
3. access to a work telephone and desktop computer with internet,
4. not pregnant,
5. no planned absence >1 week during the trial,
6. not chair-bound or uniquely impaired such that reducing occupational sitting time was not feasible,
7. no pre-existing musculoskeletal disorder.

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-12; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simon H Till, Principal Investigator — Sheffield Hallam University

REFERENCES:
- [Background] Neuhaus M, Eakin EG, Straker L, Owen N, Dunstan DW, Reid N, Healy GN. Reducing occupational sedentary time: a systematic review and meta-analysis of evidence on activity-permissive workstations. Obes Rev. 2014 Oct;15(10):822-38. doi: 10.1111/obr.12201. Epub 2014 Jul 11. PMID 25040784
- [Background] Wilmot EG, Edwardson CL, Achana FA, Davies MJ, Gorely T, Gray LJ, Khunti K, Yates T, Biddle SJ. Sedentary time in adults and the association with diabetes, cardiovascular disease and death: systematic review and meta-analysis. Diabetologia. 2012 Nov;55(11):2895-905. doi: 10.1007/s00125-012-2677-z. Epub 2012 Aug 14. PMID 22890825
- [Background] Kazi A, Duncan M, Clemes S, Haslam C. A survey of sitting time among UK employees. Occup Med (Lond). 2014 Oct;64(7):497-502. doi: 10.1093/occmed/kqu099. Epub 2014 Aug 18. PMID 25135938
- [Background] Kessler RC, Barber C, Beck A, Berglund P, Cleary PD, McKenas D, Pronk N, Simon G, Stang P, Ustun TB, Wang P. The World Health Organization Health and Work Performance Questionnaire (HPQ). J Occup Environ Med. 2003 Feb;45(2):156-74. doi: 10.1097/01.jom.0000052967.43131.51. PMID 12625231

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Office-based workplace (UK)
Groups:
- Height-adjustable Workstation: Participants received a height-adjustable workstation for four weeks
  Height-adjustable workstation
Period: Overall Study
Arm/Group | Height-adjustable Workstation | Control
Started | 22 | 9
Completed | 22 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Height-adjustable Workstation | Control | Total
Number analyzed (Participants) | 22 | 9 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 9 | 31
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (10.3) | 37 (7.26) | 43.38 (9.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 7 | 19
  Male | 10 | 2 | 12
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 22 | 9 | 31

OUTCOME MEASURES:

1. Primary Outcome: Change in Workplace Sedentary Time
Description: The amount of time a participant spends sitting whilst in the workplace (minutes). This was measured using a thigh-worn ActivPAL accelerometer.
Time Frame: Baseline (0 weeks), 4 weeks after installation of height-adjustable workstations
Measure: Mean (Standard Deviation); unit: Minutes
Groups:
- Height-adjustable Workstation: Participants that received a height-adjustable workstation
- Control: Participants that did not receive a height-adjustable workstation
Arm/Group | Height-adjustable Workstation | Control
Number analyzed (Participants) | 11 | 6
Minutes
  Baseline | 369 (43.75) | 355 (73.69)
  4-Weeks after installation | 229 (46.35) | 338 (70.4)

2. Secondary Outcome: Change in Workplace Absenteeism Using the World Health Organisation Health and Work Performance Questionnaire
Description: Self-reported absolute absenteeism (the amount of time a participant was absent from work for during the previous 7-days) measured using the World Health Organisation Health and Work Performance Questionnaire. This is calculated in relation to a participants contracted hours, therefore a negative score shows that a participant worked less than they are contracted to, where as a positive score means a participant reported working more hours than they are contracted to.
Time Frame: Baseline (0 weeks), 4 weeks after installation of height-adjustable workstations
Measure: Median (Full Range); unit: Hours worked in last 7-days
Arm/Group | Height-adjustable Workstation | Control
Number analyzed (Participants) | 21 | 7
Hours worked in last 7-days
  Baseline Absenteeism | -4 [-68 to 28] | -8 [-24 to 8]
  4-Week Absenteeism | 0 [-80 to 60] | 0 [-48 to 60]

3. Secondary Outcome: Change in Workplace Presenteeism Using the World Health Organisation Health and Work Performance Questionnaire
Description: Self-reported absolute presenteeism (an employees productivity during working hours) measured using the World Health Organisation Health and Work Performance Questionnaire. The higher the percentage, the more productive a participant felt they were. 100% means that they felt they were productive the whole time they were working. Presenteeism can be impacted upon by illness and other health conditions, if a person was feeling ill or had a back problem, this may mean that they are less productive whilst at work.
Time Frame: Baseline (0 weeks), 4 weeks after installation of height-adjustable workstations
Measure: Median (Full Range); unit: Percentage of job able to perform
Groups:
- Height-adjustable Workstation: Participants received a height-adjustable workstation
- Control: Participants that did not received a height-adjustable workstation
Arm/Group | Height-adjustable Workstation | Control
Number analyzed (Participants) | 21 | 7
Percentage of job able to perform
  Baseline Presenteeism | 80 [40 to 100] | 80 [60 to 90]
  4-Week Presenteeism | 80 [50 to 100] | 90 [70 to 100]

ADVERSE EVENTS:
Arm/Group | Height-adjustable Workstation | Control
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/9
Other Adverse Events (participants affected / at risk) | 0/22 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes